CLINICAL TRIAL: NCT06704204
Title: Long-acting Injectable Antiretroviral Treatment to Improve HIV Treatment Among Justice-involved Persons Being Released to the Community (Study #3; Aim 2 Injectable CAB/RPV Pilot)
Brief Title: Long-acting Injectable Antiretroviral Treatment to Improve HIV Treatment Among Justice-involved Persons Being Released to the Community
Status: Not yet recruiting | Type: Observational
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Curt Beckwith, Professor of Medicine, The Miriam Hospital
Other Study IDs: 20241441; R34DA057165 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: HIV
Keywords: HIV infection; substance use disorders; community re-entry; HIV treatment; long-acting injectable; incarceration
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — cabotegravir; Rilpivirine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- people with HIV (PWH) who are experiencing community re-entry: ART is highly effective in controlling HIV and can significantly reduce HIV transmission when viral suppression is achieved. ART is usually administered as a combination of antiretroviral medications taken orally daily. Despite the convenience of single pill fixed-dose ART regimens, many persons, including justice involved substance users, struggle with daily ART adherence and consequently experience disease progression, emergence of HIV resistance, and contribute to HIV transmission. Long-acting injectable (LAI) ART is a new alternative to help overcome the challenges of adhering to daily pills. LAI ART is administered by intramuscular injection every four weeks and the first LAI regimen, cabotegravir (CAB) combined with rilpivirine (RPV), was FDA-approved in January 2021 for treatment of HIV infection. While rollout of LAI ART has recently begun, using LAI ART among PWH during the challenging community re-entry period has the substantial potential to improve HIV treatment outcomes.
  Interventions: Drug: The first FDA-approved LAI ART regimen includes an integrase inhibitor, cabotegravir (CAB), and a non-nucleoside reverse transcriptase inhibitor, rilpivirine (RPV) combined 4 wks

INTERVENTIONS:
Drug: The first FDA-approved LAI ART regimen includes an integrase inhibitor, cabotegravir (CAB), and a non-nucleoside reverse transcriptase inhibitor, rilpivirine (RPV) combined 4 wks — To date, there have been no studies looking at the use of LAI ART among justice involved PWH, yet a significant opportunity exists to improve HIV treatment outcomes in this high risk population.30

SUMMARY:
The federal research award entitles "Long-acting injectable antiretroviral treatment to improve HIV treatment among justice-involved persons being released to the community" aims to Conduct interviews with justice and treatment experienced PWH (n=20), and carceral and community key stakeholders (n=20), to obtain guidance on the development and implementation of a protocol to transition PWH with viral suppression on oral ART to LAI ART in prison with continuation during community re-entry; develop an initial LAI ART community re-entry protocol based on Aim 1 findings and conduct an open label pilot study. Post-release follow up will occur for three months among 20-30 incarcerated PWH eligible for LAI ART who are near release from prison in order to optimize protocol procedures including participant recruitment, initiation of LAI ART in prison, transition of LAI ART to community providers, and to pilot study retention methods and assessments, including post-release HIV viral loads and urine drug testing, during the follow-up period.

DETAILED DESCRIPTION:
R34-funded mixed methods study that will develop and pilot test an LAI ART protocol designed specifically for PWH who are experiencing community re-entry

ELIGIBILITY:
Inclusion Criteria:

* 1) ≥18 years of age; 2) English speaking; 3) HIV positive (confirmed by medical record review); 4) receiving oral ART; 5) documentation of HIV viral suppression (< 50 copies/mL) on oral ART within 12 weeks of recruitment; 5) eligible to transition from oral ART to injectable CAB/RPV based upon medical record review and pre-treatment evaluation; 6) willing to transition ART to injectable CAB/RPV; 7) anticipated release from MDPSCS facility within 12 weeks; 8) anticipated release to Baltimore City; 9) willing to receive post-release CAB/RPV injections at community-based sites; and 10) able to provide informed consent for study participation.

Exclusion Criteria:

* Persons who are currently prescribed injectable CAB/RPV within MDPSCS will not be eligible for study enrollment, however, we do not anticipate use of injectable CAB/RPV will be common in this population during the conduct of this study given slow roll out in the community to date and no experience within carceral facilities. Potential participants unable to provide informed consent, including people with severe mental illness (e.g., untreated psychosis, bipolar disorder with mania; adequately treated psychiatric disorders and appropriate psychotropic medications will be allowed) requiring immediate treatment or with mental illness limiting their ability to participate (e.g., dementia), will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from participating carceral settings through direct referral from carceral HIV providers. We will plan to enroll women and men for the open label pilot study to ensure we gain experience with recruitment from facilities for both women and men. In addition, recruitment of women study participants at this stage will be important given additional eligibility requirements for women being considered for injectable CAB/RPV (pregnancy considerations following release).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Viral Suppression Out of Total Participants | 3 months
  HIV viral load

SECONDARY OUTCOMES:
Number of Participants with Adherence Out of Total Participants | 3 months
  adherence to LAI ART medication
Number of Participants Retention Out of Total Participants | 3 months
  Loss to follow up (LTFU)

CONTACTS AND LOCATIONS:
Overall Officials: Curt G Beckwith, MD, Principal Investigator — The Miriam Hospital

IPD SHARING:
Plan to Share IPD: No
Study population are vulnerable population, including people with HIV (PWH) and incarcerated individuals.